CLINICAL TRIAL: NCT03452579
Title: CA209-382 A Randomized Phase 2 Open Label Study of Nivolumab Plus Standard Dose Bevacizumab Versus Nivolumab Plus Low Dose Bevacizumab in Recurrent Glioblastoma (GBM)
Brief Title: Nivolumab Plus Standard Dose Bevacizumab Versus Nivolumab Plus Low Dose Bevacizumab in GBM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Peereboom (Other)
Responsible Party: Sponsor-Investigator, David Peereboom, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1317
Record Dates: First submitted 2018-01-29; First posted 2018-03-02 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
Keywords: Nivolumab; Bevacizumab
MeSH Terms: conditions — Glioblastoma | interventions — Nivolumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab + Standard Dose Bevacizumab (Active Comparator): nivolumab 240 mg IV and standard dose bevacizumab 10 mg/kg every 2 weeks until disease progression or unacceptable toxicity.
  Nivolumab is to be administered first. The second infusion will be bevacizumab, and will start no sooner than 10 minutes after completion of the nivolumab infusion
  Interventions: Drug: Nivolumab; Drug: Standard Dose Bevacizumab
- Nivolumab + Low Dose Bevacizumab (Experimental): nivolumab 240 mg IV and low dose bevacizumab 3mg/kg every 2 weeks until disease progression or unacceptable toxicity
  Nivolumab is to be administered first. The second infusion will be bevacizumab, and will start no sooner than 10 minutes after completion of the nivolumab infusion
  Interventions: Drug: Nivolumab; Drug: Low Dose Bevacizumab

INTERVENTIONS:
Drug: Nivolumab — 240mg
  Other Names: Opdivo
Drug: Standard Dose Bevacizumab — 10mg/kg
  Other Names: Avastin
  Arms: Nivolumab + Standard Dose Bevacizumab
Drug: Low Dose Bevacizumab — 3mg/kg
  Other Names: Avastin
  Arms: Nivolumab + Low Dose Bevacizumab

SUMMARY:
The purpose of this study is to test the effectiveness (how well the drug works), safety and tolerability of an investigational drug called nivolumab (also known as BMS-936558) in glioblastoma (a malignant tumor, or GBM), when added to bevacizumab.

Nivolumab is an antibody (a kind of human protein) that is being tested to see if it will allow the body's immune system to work against glioblastoma tumors. Opdivo (nivolumab ) is currently FDA approved in the United States for melanoma (a type of skin cancer), non-small cell lung cancer, renal cell cancer (a type of kidney cancer), Hodgkin's lymphoma but is not approved in glioblastoma. nivolumab may help your immune system detect and attack cancer cells.

Bevacizumab is a drug which works on the blood vessel that supply the tumor and potentially can starve the tumor by cutting off the blood supply to these tumors. Bevacizumab is commercially available and FDA approved for individuals with recurrent glioblastoma.

This study has two study groups. Arm 1 will receive the study drug nivolumab 240mg and bevacizumab 10 mg (standard dose) every 2 weeks and Arm 2 will receive the study drug nivolumab 240 mg and bevacizumab 3 mg (low dose) every 2 weeks. A process will be used to assign participants, by chance, to one of the study groups. Neither participants nor doctors can choose which group participants are in. This is done by chance because no one knows if one study group is better or worse than the other. 90 total participants are expected to participate in this study (45 participants in each arm).

Your total participation in this study from the time you have signed the informed consent to your last visit, including follow-up visits, may be more than three years (depending on what effect the treatment has on your cancer, and how well you tolerate the treatment).

DETAILED DESCRIPTION:
Primary Endpoint(s)

-To evaluate the efficacy of nivolumab when administered with standard and low bevacizumab dosing among recurrent glioblastoma patients as measured by the rate of overall survival at twelve months.

Secondary Endpoint(s)

* To evaluate the safety and tolerability of nivolumab in combination with bevacizumab administered according to standard and low dosage schedules for recurrent glioblastoma patients.
* To compare progression free survival (PFS) at 6 months of nivolumab when administered with standard and low bevacizumab dosing for recurrent glioblastoma patients.
* To compare the overall survival rate of nivolumab when administered with standard and low bevacizumab dosing for recurrent glioblastoma patients.
* To compare progression free survival (PFS) of when administered with standard and low bevacizumab dosing for recurrent glioblastoma patients.
* To compare the objective response rate (ORR) of nivolumab and bevacizumab administered according to standard and low dosage schedules for recurrent glioblastoma patients

Study design and duration: This is a randomized, open-label, phase 2 safety study of nivolumab and bevacizumab administered according to standard and low dosage schedules in adult (≥ 18 years) participants with a first recurrence or second recurrence of glioblastoma (GBM). Participants must have received previous treatment with radiotherapy and one recurrence. The study will allow participants that require decadron up to 4mg/day to participate. Participants will undergo 1:1 randomization to receive treatment with either nivolumab (240 mg flat dosing IV every 2 weeks) and bevacizumab administered according to standard (10 mg/kg IV every 2 weeks; Arm A) and low (3 mg/kg IV every 2 weeks; Arm B) dosage schedules for recurrent glioblastoma participants. The study will allow participants that require decadron up to 4 mg/ day to participate in the study.

Note - In view of the Covid 19 crisis, all in person visits can be substituted for virtual visit. All nursing toxicity checks can be performed over the phone rather than in person

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by MRI.
* Histologically confirmed diagnosis of supratentorial glioblastoma
* Previous first line treatment with at least radiotherapy
* Documented first recurrence of GBM by diagnostic biopsy or contrast enhanced magnetic resonance imaging (MRI) performed within 21 days of randomization per RANO criteria.
* If first recurrence of GBM is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either:

  * histopathologic confirmation of recurrent tumor, or
  * new enhancement on MRI outside of the radiotherapy treatment field
* An interval of > 28 days and full recovery (i.e., no ongoing safety issues) from surgical resection prior to randomization.
* Karnofsky performance status (KPS) of 70 or higher (Appendix 1)
* Life expectancy > 12 weeks
* Up to ten unstained slides of 5 microns thickness or a block of tissue will be required to be sent if tissue is available. If the tissue is not available then Principal investigator permissions is required prior to enrollment
* Women of childbearing potential (WOCBP,) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 1 day prior to the start of study drug
* Women must not be breastfeeding
* WOCBP must use appropriate method(s) of contraception from the time of enrollment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 6 months post treatment completion for a treatment arm A (nivolumab + standard dose bevacizumab)and treatment arm B (nivolumab + low dose bevacizumab).
* Men who are sexually active with WOCBP must use contraceptive method such as male condom with spermicide. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion.
* Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception.
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements.
* Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly.
* At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:
* HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

  * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena® by WOCBP subjects or male subject's WOCBP partner.
  * Nonhormonal IUDs, such as ParaGard
  * Tubal ligation
  * Vasectomy.
  * Complete Abstinence* ---*Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence.
* LESS EFFECTIVE METHODS OF CONTRACEPTION

  * Diaphragm with spermicide
  * Cervical cap with spermicide
  * Vaginal sponge
  * Male Condom without spermicide*
  * Progestin only pills by WOCBP subjects or male subject's WOCBP partner
  * Female Condom* ---*A male and female condom must not be used together
* Women of Child Bearing Potential (WOCBP)

  --A women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, women under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40mIU/mL to confirm menopause.*

  ---*Women treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgment in checking serum FSH levels. If the serum FSH level is > 40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal:
  * 1 week minimum for vaginal hormonal products (rings, creams, gels)
  * 4 week minimum for transdermal products
  * 8 week minimum for oral products
* Other parenteral products may require washout periods as long as 6 months Each of the criteria in the checklist that follows must be met in order for a patient to be considered eligible for this study. Use the checklist to confirm a patient's eligibility. The checklist must be completed for each patient and must be signed and dated by the treating physician.
* Recovery from the toxic effects of prior therapy, with a minimum time of:

  * (≥) 28 days elapsed from the administration of any investigational agent
  * (≥) 28 days elapsed from the administration of any prior cytotoxic agents, except
  * (≥)14 days from vincristine, ≥ 21 days from procarbazine, and ≥ 42 days from
  * nitrosureas
  * (≥) 14 days elapsed from administration of any non-cytotoxic agent (e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid)
* Screening/Baseline laboratory values must meet the following criteria (using CTCAE v5.0):

  * WBC ≥ 2000/uL
  * Neutrophils ≥ 1500/uL
  * Platelets ≥ 100x103/uL
  * Hemoglobin ≥ 9.0 g/dL
  * Serum creatinine < 1.5 x ULN or creatinine clearance (CrCl) > 40 mL/min (using the Cockcroft-Gault formula)

    * Female CrCl = (140 - age in years) x weight in kg x 0.85 /72 x serum creatinine in mg/dL
    * Male CrCl = (140 - age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL
  * AST ≤ 3x ULN
  * ALT≤ 3x ULN
  * Pregnancy test (serum)
  * Bilirubin ≤ 1.5x ULN (except subjects with Gilbert Syndrome, who can have
  * Total bilirubin < 3.0 mg/dL)

Exclusion Criteria:

* More than two recurrences of GBM
* Presence of extracranial metastatic, significant leptomeningeal disease or tumors primarily localized to the brainstem or spinal cord.
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic and systemic immunosuppressive treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects have any other condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent are permitted in absence of active autoimmune disease
* Previous radiation therapy with anything other than standard radiation therapy (i.e., focally directed radiation) administered as first line therapy.
* Previous treatment with carmustine wafer except when administered as first line treatment and at least 6 months prior to randomization
* Previous bevacizumab or other VEGF or anti-angiogenic treatment
* Previous treatment with a PD-1, PD-L1 or CTLA-4 targeted therapy
* Evidence of > Grade 1 CNS hemorrhage on the baseline MRI scan
* Inadequately controlled hypertension (defined as systolic blood pressure ≥160 mmHg and /or diastolic blood pressure ≥100 mmHg) within 7 days of first study treatment
* Prior history of hypertensive crisis, hypertensive encephalopathy, reversible posterior leukoencephalopathy syndrome (RPLS);
* Prior history of gastrointestinal diverticulitis, perforation, or abscess;
* Clinically significant (i.e., active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment;
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism ≥ NCI CTCAE Grade 3 within 3 months prior to start of study treatment;
* History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month prior to randomization;
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation);
* Current or recent (within 10 days of study enrollment) use of anticoagulants that, in the opinion of the investigator, would place the subject at significant risk for bleeding. Prophylactic use of anticoagulants is allowed;
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study;
* Minor surgical procedure (e.g., stereotactic biopsy within 7 days of first study treatment; placement of a vascular access device within 2 days of first study treatment);
* History of intracranial abscess within 6 months prior to randomization;
* History of active gastrointestinal bleeding within 6 months prior to randomization;
* Serious, non-healing wound, active ulcer, or untreated bone fracture;
* Subjects unable (due to existent medical condition, e.g., pacemaker or ICD device) or unwilling to have a head contrast enhanced MRI
* Positive test for hepatitis B virus surface antigen (HBV sAg) or detectable hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* History of severe hypersensitivity reaction to any monoclonal antibody
* Patients that require decadron > 4 mg/ day or equivalent of steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2025-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] de Melo SM, Elias Nunes da Silva ME, Torloni MR, Riera R, De Cicco K, Latorraca CO, Pinto ACPN. Anti-PD-1 and anti-PD-L1 antibodies for glioma. Cochrane Database Syst Rev. 2025 Jan 8;1(1):CD012532. doi: 10.1002/14651858.CD012532.pub2. PMID 39777725

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Standard Dose Bevacizumab: nivolumab 240 mg IV and standard dose bevacizumab 10 mg/kg every 2 weeks until disease progression or unacceptable toxicity.
  Nivolumab is to be administered first. The second infusion will be bevacizumab, and will start no sooner than 10 minutes after completion of the nivolumab infusion
  Nivolumab: 240mg
  Standard Dose Bevacizumab: 10mg/kg
- Nivolumab + Low Dose Bevacizumab: nivolumab 240 mg IV and low dose bevacizumab 3mg/kg every 2 weeks until disease progression or unacceptable toxicity
  Nivolumab is to be administered first. The second infusion will be bevacizumab, and will start no sooner than 10 minutes after completion of the nivolumab infusion
  Nivolumab: 240mg
  Low Dose Bevacizumab: 3mg/kg
Period: Overall Study
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Started | 45 | 45
Completed | 3 | 2
Not Completed | 42 | 43
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Disease progression, relapse during active treatment | 38 | 37
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Full Range); unit: Years] | 60.7 [27.4 to 81.0] | 60.5 [27.7 to 86.4] | 60.6 [27.4 to 86.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 32 | 29 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 43 | 86
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 40 | 42 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90
Baseline Karnofsky Performance Scale (KPS) [Count of Participants; unit: Participants] — KPS Index allows participants to be classified as to their functional impairment. Scores range from 0% to 100%. The lower the Karnofsky score, the worse the survival for most serious illnesses.
  Participants
    70% | 11 | 13 | 24
    80% | 18 | 17 | 35
    90% | 15 | 13 | 28
    100% | 0 | 1 | 1
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 12 Months (OS-12)
Description: OS-12 is the percentage of participants in the analysis population who remain alive for at least twelve months following initiation of study therapy.
  Participants without efficacy evaluation data or without survival data will be censored at Day 1
Time Frame: Up to 12 months after beginning therapy
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
Percentage of participants | 41.1 [26.1 to 56.1] | 37.7 [23.1 to 52.4]

2. Secondary Outcome: Progression-Free Survival (PFS) at Six Months
Description: The percentage of participants in the analysis population who remain progression-free for at least six months following initiation of study therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
  Participants without efficacy evaluation data or without survival data will be censored at Day 1
Time Frame: Up to six months after beginning treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
Percentage of participants | 46.7 [32.1 to 61.2] | 44.6 [29.4 to 59.8]

3. Secondary Outcome: Overall Survival (OS)
Description: OS, as defined as number of participants alive from beginning of treatment up to 6 six months
  Participants without efficacy evaluation data or without survival data will be censored at Day 1
Time Frame: Up to six months after beginning treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
Percentage of participants | 75.1 [62.3 to 87.9] | 57.4 [42.9 to 71.9]

4. Secondary Outcome: Overall Survival (OS)
Description: OS, as defined as the percentage of participants alive from beginning of treatment up to 18 months.
  Participants without efficacy evaluation data or without survival data will be censored at Day 1
Time Frame: Up to 18 months after beginning treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
Percentage of participants | 30.9 [15.7 to 46.1] | 22.5 [8.5 to 36.5]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Proportion of participants in the analysis population who have complete response (CR) or partial response (PR) using Radiologic Assessment in Neuro-Oncology criteria (RANO) criteria.
  Participants without efficacy evalaluation data or survival data censored at day 1. Participants without measurable disease will not be included.
Time Frame: Up to 3 years after beginning treatment
Measure: Number; unit: percentage of participants
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
percentage of participants | 18 | 16

6. Secondary Outcome: Progression-Free Survival
Description: Median time from allocation to first documented disease progression per RANO or death due to any cause, whichever occurs first. Those without efficacy eval. data or survival data censored at day 1
  RANO - progressive disease:
  * (>) 25% increase in sum of products of perpendicular diameters of measurable lesions (over best response [smallest tumor size] or baseline if no decrease) on stable/increasing corticosteroid doses
  * Any new measurable lesion that when added to change in initial tumor(s) exceeds 25% increase in x-sectional area.
  * Clear clinical deterioration not attributable to causes apart from tumor. Def. is left to discretion of PI but recommended is: Decline in KPS from 100 or 90 to <= 70, decline in KPS of at least 20 from <= 80, or decline in KPS from any baseline to <= 50, for >= 7 days, be considered neurologic deterioration, unless attributable to co-morbid events or changes in corticosteroid dose.
  * Failure to return for eval. due to death or deteriorating condition
Time Frame: Up to 3 years after beginning treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
months | 4.1 [3.2 to 7.0] | 5.6 [3.7 to 6.8]

7. Secondary Outcome: Duration of Response
Description: Time from first RANO response to disease progression in participants who achieve a PR or better
  Participants without efficacy evaluation data or without survival data will be censored at Day 1
Time Frame: Up to 3 years after beginning treatment
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
Number analyzed (Participants) | 45 | 45
months | 5.2 [3.5 to 6.6] | 5.2 [3.4 to 6.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were on study up to 3 years
Arm/Group | Nivolumab + Standard Dose Bevacizumab | Nivolumab + Low Dose Bevacizumab
All-Cause Mortality (participants affected / at risk) | 37/45 | 40/45
Serious Adverse Events (participants affected / at risk) | 25/45 | 21/45
Other Adverse Events (participants affected / at risk) | 45/45 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Standard Dose Bevacizumab (N=45) | Nivolumab + Low Dose Bevacizumab (N=45)
ALT Increase (Blood and lymphatic system disorders) | 1 | 1
Neutrophil decreased (Blood and lymphatic system disorders) | 1 | 1
Deep vein thrombosis (Cardiac disorders) | 3 | 2
Hypertension (Cardiac disorders) | 4 | 3
Pulmonary Embolism (Cardiac disorders) | 3 | 2
Fatigue (General disorders) | 6 | 1
Infection (General disorders) | 3 | 1
Pain (General disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Liver Function Abnormal (Gastrointestinal disorders) | 2 | 0
Abnormal Electrolytes (Investigations) | 1 | 0
Immune System Other Cerebrit (Investigations) | 0 | 1
Lipase Increase (Investigations) | 2 | 0
Serum Amylase Increased (Investigations) | 1 | 0
Gait Imbalance (Musculoskeletal and connective tissue disorders) | 3 | 3
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 7 | 4
Headaches (Nervous system disorders) | 3 | 0
Intracranial Hemorrhage (Nervous system disorders) | 1 | 1
Other Neurologic (Nervous system disorders) | 2 | 5
Seizure (Nervous system disorders) | 3 | 3
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1
Upper Resipratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
CPK Increased (Renal and urinary disorders) | 1 | 0
Cognitive (Nervous system disorders) | 4 | 1
Aphasia (Nervous system disorders) | 1 | 1
Hyperglycemia (Investigations) | 2 | 0
Abnormal LFT (Gastrointestinal disorders) | 2 | 0
Dehydration (General disorders) | 0 | 1
Lethargy (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Standard Dose Bevacizumab (N=45) | Nivolumab + Low Dose Bevacizumab (N=45)
ALT increased (Blood and lymphatic system disorders) | 11 | 8
Bleed (Blood and lymphatic system disorders) | 13 | 8
Platelet count decreased (Blood and lymphatic system disorders) | 12 | 9
Hypertension (Cardiac disorders) | 15 | 7
Fatigue (General disorders) | 29 | 19
Diarrhea (Gastrointestinal disorders) | 17 | 12
Nausea (Gastrointestinal disorders) | 10 | 11
AST increased (Investigations) | 9 | 5
Hypothroidism (Investigations) | 5 | 6
Lipase Increased (Investigations) | 14 | 6
Serum amylase increased (Investigations) | 9 | 4
Body pain/stiffness (Musculoskeletal and connective tissue disorders) | 13 | 11
Joint Pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Headache (Nervous system disorders) | 20 | 12
Other-neurologic (Nervous system disorders) | 13 | 12
Proteinuria (Renal and urinary disorders) | 15 | 17
Hiccups/hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 12 | 8
Seizure (Nervous system disorders) | 14 | 13
Behavioral Side effect (Nervous system disorders) | 8 | 10
Chest Pain (Cardiac disorders) | 7 | 1
Eye Discomfort (Eye disorders) | 3 | 5
Cough (General disorders) | 8 | 10
Flu Symptoms (General disorders) | 12 | 13
Infection (General disorders) | 9 | 7
Insomnia (General disorders) | 6 | 2
Weight loss (General disorders) | 6 | 7
Abdominal Discomfort (Gastrointestinal disorders) | 7 | 2
Constipation (Gastrointestinal disorders) | 4 | 9
Dysphagia (Gastrointestinal disorders) | 4 | 6
Vomiting (Gastrointestinal disorders) | 4 | 7
Abnormal Electrocytes (Investigations) | 18 | 15
Hyperglycemia (Investigations) | 12 | 8
General Muscle Weakness (Investigations) | 12 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT03452579/Prot_SAP_002.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03452579/ICF_001.pdf